CLINICAL TRIAL: NCT01073085
Title: Effectiveness of a French Automated Web-based Smoking Cessation Program : a Randomized Controlled Trial
Brief Title: Effectiveness of a French Automated Web-based Smoking Cessation Program
Acronym: Stamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut national de prevention et d'education pour la sante (Other Government)
Responsible Party: Principal Investigator, Dr. Pierre Arwidson, Directeur des affaires scientifiques, Institut national de prevention et d'education pour la sante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Stamp
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Tobacco Consumption
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based coaching (Experimental): Those in the "coaching" arm will benefit from e-mails with advice, information, support for smoking cessation. These mails will be adapted to their personal profile.
  Interventions: Behavioral: Web-based automated "coaching" by e-mails
- Self-help guide (Active Comparator): Those in the "active comparator arm" will be allowed to download a self-help guide with step-by-step advice for smoking cessation.
  Interventions: Behavioral: Self-help guide

INTERVENTIONS:
Behavioral: Web-based automated "coaching" by e-mails
  Arms: Web-based coaching
Behavioral: Self-help guide
  Arms: Self-help guide

SUMMARY:
The purpose of this study is to investigate the effectiveness of a French fully automated web-based smoking cessation program known as the "coaching", by comparing it to an online self-help guide.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Smoker
* Willing to quit smoking in the next two weeks
* Having a regular access to Internet
* Having a personal e-mail address
* Not having benefited from the "coaching" the investigators want to assess yet

Exclusion Criteria:

* No personal e-mail address
* Not able to give the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2478 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage of abstinent people between the two arms of the trial, 6 months after inclusion | 6 months after inclusion
  The investigators will compare the percentage of smokers who successfully quit, 6 months after their inclusion in the study. Point prevalence abstinence will be measured (not smoking, event a puff, in the week preceding the questioning).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Arwidson, Doctor, Study Director — Institut national de prevention et d'education pour la sante
Locations (1):
- Institut national de prevention et d'education pour la sante, Saint-Denis, France